CLINICAL TRIAL: NCT01232868
Title: Systems Biology of Trivalent Influenza Vaccine (TIV) in Young and Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nadine Rouphael, MD, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00046787; NIH (Other: NIH U19 AI 90023); VAX-001 (Other: Other)
Record Dates: First submitted 2010-10-23; First posted 2010-11-02 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: Innate immunity; Adaptive immunity; Slu shot; Elderly
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Age 25-40 (Other): Trivalent Influenza vaccine given to age 25-40
  Interventions: Biological: trivalent Influenza vaccine (TIV)
- Age ≥65 (Other): Trivalent Influenza vaccine given to age≥65
  Interventions: Biological: trivalent Influenza vaccine (TIV)

INTERVENTIONS:
Biological: trivalent Influenza vaccine (TIV) — 0.5 ml IM as a single dose in a prefilled syringe.
  Other Names: Fluzone

SUMMARY:
Vaccination is the most effective way of preventing infectious diseases. Despite the success of vaccines in general, vaccines induce diminished antibody responses and lower protection in the elderly in particular. This could be explained by a defect in the early responses of an ageing immune system. A better understanding of the basic immunological mechanisms that mediate vaccine efficacy is incomplete. Such information is critical and could greatly decrease both the cost and the time to new vaccine development particularly for the geriatric population.

In this trial, the investigators will study the immunologic differences of an FDA approved licensed influenza vaccine between a younger and an older group. Twenty two healthy volunteers between the age of 25-40 and forty four healthy volunteers above the age of 65 will be enrolled in the study. Each participant in the study will be given one flu shot. Blood work will be obtained prior to vaccination, one day, three days, seven days, fourteen days, as well as one month and six months after vaccination. Throughout the duration of the study, the participants will be monitored for safety.

DETAILED DESCRIPTION:
RATIONALE:Trivalent Influenza vaccine (TIV) is known to induce diminished functional antibody responses and lower protection in the elderly. Here we hypothesize that this is due to intrinsic defects in innate responses which translates into suboptimal Hemagglutination Inhibition Assay (HAI) titers. Therefore, early innate signatures of vaccination should correlate with, and predict the immunogenicity of TIV in the young and elderly.

STUDY DESIGN: Single center, open label study in which adult healthy volunteers with no contraindications to immunization will be vaccinated with TIV. Blood samples will be collected on Days D0 (at enrollment) and D1, D3, D7, D14, D30, D180 post vaccination to study innate and/or adaptive immunity markers. Even though influenza vaccination is considered safe, volunteers will be asked to report any local or systemic adverse events (AEs) from Day 0 (vaccination) to Day 7 in memory aids. Reactogenicity events will also be evaluated by injection site examination on visits at D0, D1, D3 and D7. Volunteers will be also asked to report local and systemic AEs developing the day of a blood draw.

Additionally, only AEs considered related (unlikely, possibly, probably or definitely related) will be collected and reported in this study from Day 0 (vaccination) to Day 180. After Day 30 only related SAEs will be collected and reported.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals aged 25-40 years, or ≥65 years old.
2. Able to understand and give informed consent.
3. Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for ≥1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods for 30 days before and 30 days after trivalent Influenza vaccination.

Exclusion Criteria:

1. Receipt of immune products:

   * Receipt of blood products 3 months prior to study entry or expected receipt through 6 months after study entry
   * Receipt of any live virus vaccines within 4 weeks prior to study entry or expected receipt within 4 weeks after study entry*
   * Receipt of any inactivated vaccine within 2 weeks or expected receipt within 2 weeks after study entry*
   * Receipt of the 2010-2011 influenza vaccine
2. Documented influenza infection during the 2010-2011 influenza season. Not excluded from the study, volunteers with prior upper respiratory infections during the 2010-2011 influenza illness.
3. Presence of co-morbidities or immunosuppressive states such as:

   * Chronic medical problems including (but not limited to) insulin dependent diabetes, severe heart disease, severe lung disease, severe liver disease, severe kidney disease, auto immune diseases, severe gastrointestinal diseases, and uncontrolled hypertension.
   * Alcohol or drug abuse and psychiatric conditions that in the opinion of the investigator would preclude compliance with the trial or interpretation of safety or endpoint data.
   * Impaired immune function or chronic infections including (but not limited to) HIV, hepatitis B or C; organ transplant; cancer; current and/or expected receipt of chemotherapy, radiation therapy or any other cytotoxic or immunosuppressive therapy [i.e. more than 10 mg of prednisone given daily or on alternative days for 2 weeks or more in the past 3 months*; receipt of high-dose inhaled steroids is also an exclusion criteria (nasal and topical steroids are allowed.)], congenital immunodeficiency, anatomical or functional asplenia.
   * Pregnancy or breast feeding
4. Conditions that could affect the safety of the volunteers such as:

   * Severe reactions to prior vaccination with TIV, including anaphylaxis.
   * History of Guillain Barré syndrome
   * History of bleeding disorders
   * Any allergy to any component of the vaccine including egg allergy.
5. Volunteers with any acute illness, including any fever (> 100.4 F [> 38.0C], regardless of the route) within 3 days prior to study entry *.
6. Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.

   * Note:

An individual who initially is excluded from study participation based on one or more of the time-limited exclusion criteria (e.g., acute illness, receipt or expected receipt of live or inactivated vaccines ) may be reconsidered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria.

Subjects receiving > 10 mg/day of prednisone or its equivalent daily or on alternate days for more than 2 weeks may enter the study after therapy has been discontinued for more than 3 months.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (1):
- Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Atlanta Metropolitan Area 2010-2011
Pre-assignment Details: There were 4 screen failures :
  * one unable to obtain blood pre-vaccination
  * two with elevated blood pressure readings
  * one with progressive medical illness
Groups:
- Age 25-40 Years: Healthy participants between the ages of 25 to 40 years of age received 0.5 ml of the trivalent Influenza vaccine (TIV) administered via the intramuscular route in the deltoid muscle as a single dose.
- Age ≥65 Years: Healthy participants 65 years or older received 0.5 ml of the trivalent Influenza vaccine (TIV) administered via the intramuscular route in the deltoid muscle as a single dose.
Period: Overall Study
Arm/Group | Age 25-40 Years | Age ≥65 Years
Started | 22 | 44
Completed | 20 | 40
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Population: All subjects received a single dose of the trivalent Influenza vaccine (TIV).
Groups:
- Age ≥65 Years: Healthy participants 65 years and older received 0.5 ml of the trivalent Influenza vaccine (TIV) administered via the intramuscular route in the deltoid muscle as a single dose.
- Total: Total of all reporting groups
Arm/Group | Age 25-40 Years | Age ≥65 Years | Total
Number analyzed (Participants) | 22 | 44 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 0 | 22
  >=65 years | 0 | 44 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 23 | 37
  Male | 8 | 21 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 20 | 41 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 12 | 40 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 44 | 66

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, Measured by the Number of Subjects With a Change in Innate Immune Signatures
Description: The number of subjects with a change in innate immunity signatures correlating with the level of antibodies was recorded. The innate immune signatures were assessed by Fluorescence Activated Cell Sorting (FACS)/Luminex assays. The levels of antibodies to the influenza virus prior to TIV (trivalent influenza vaccine) administration and on Day 180 after receiving TIV was assessed and the number of subjects who exhibited an increase in the antibodies and, therefore, a change in their innate immune signatures, was recorded.
Time Frame: Day 0 (prior to TIV administration), Day 180 (from the time of of TIV administration)
Measure: Number; unit: participants
Arm/Group | Age 25-40 Years | Age ≥65 Years
Number analyzed (Participants) | 22 | 44
participants | 22 | 44

2. Secondary Outcome: Number of Participants With Specific B Cell Responses That Correlate With the Innate Immune Signatures
Description: The secondary outcomes will identify the number of participants with a positive B cell response to the flu shot particulary looking for antibody responses, presence of plasmablasts, antibody repertoire.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Age 25-40 Years | Age ≥65 Years
Number analyzed (Participants) | 22 | 44
participants | 21 | 40

ADVERSE EVENTS:
Time Frame: 6 months
Description: Reactogenecity for 7 days post vaccination AE for 30 days SAE for 180 days (None of the SAE were related to the vaccine-One participant had choliangiocarcinoma and bacteremia and multiorgan failure and died 6 months after receiving TIV- another SAE was in a participant with hospitalization for small bowel obstruction with complete recovery)
Arm/Group | Age 25-40 Years | Age ≥65 Years
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/44
Other Adverse Events (participants affected / at risk) | 14/22 | 29/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 25-40 Years (N=22) | Age ≥65 Years (N=44)
Cholangiocarcinoma (Hepatobiliary disorders) | 0 (0) | 1 (1) — treated with radiofrequency ablation
Multiorgan Failure (Endocrine disorders) | 0 (0) | 1 (1) — Multiorgan failure including thyroid storm
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) — No Mass no Cancer
Death (Infections and infestations) | 0 (0) | 1 (1) — E.coli bacteremia resulting in multiorgan failure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 25-40 Years (N=22) | Age ≥65 Years (N=44)
Bruise (Blood and lymphatic system disorders) | 2 (2) | 9 (9) — Bruise at phlebotomy site
Induration/Swelling (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) — Induration/Swelling at injection site in the first 7 days post vaccination
Tenderness (Skin and subcutaneous tissue disorders) | 10 (10) | 21 (21) — Tenderness at injection site in the first 7 days post vaccination
Headache (Nervous system disorders) | 3 (3) | 7 (7) — Headache in the first 7 days post vaccination
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (6) — Nausea in the first 7 days post vaccination

LIMITATIONS AND CAVEATS:
Long period of time required for detailed analysis of gene expressions in different participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No